CLINICAL TRIAL: NCT06048445
Title: Placement of Biliary Drainage Stent to Prevent Biliary Intestinal Anastomosis After Liver Transplantation in Children: A Prospective Study
Brief Title: Placement of Biliary Drainage Stent to Prevent Biliary Intestinal Anastomosis After Liver Transplantation in Children
Status: Recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weili Wang, Deputy Director of the Department, Zhejiang University
Other Study IDs: BDSPBIAP
Record Dates: First submitted 2023-09-09; First posted 2023-09-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biliary Drainage Stent group: placement of Biliary Drainage Stent in pediatric liver transplantation
  Interventions: Device: intraoperative plancement of Biliary Drainage Stent
- no Biliary Drainage Stent group: no placement of Biliary Drainage Stent in pediatric liver transplantation

INTERVENTIONS:
Device: intraoperative plancement of Biliary Drainage Stent — plancement of Biliary Drainage Stent in liver transplantation of pediatric patients
  Groups: Biliary Drainage Stent group

SUMMARY:
Liver transplantation is an effective method for treating end-stage liver disease and metabolic diseases in children. With the advancement of surgical techniques and the improvement of perioperative management, the survival rates of patients and grafts after liver transplantation have significantly improved. However, the complication of biliary stenosis after transplantation is as high as 7.3% -33.3%, and in severe cases, it can even lead to graft failure and patient death. Therefore, the occurrence of biliary stenosis after liver transplantation seriously affects the quality of life of children, increases the economic burden on families, and urgently needs to find effective methods to reduce the occurrence of this complication.

Based on the clinical practice of our center, we believe that the placement of biliary external drainage stents has the following advantages: 1 Reduce intrahepatic biliary pressure and reduce the occurrence of postoperative biliary fistula; 2. The stent has a supporting effect and can maintain the open state of the bile duct; 3. By external drainage, the quality of bile secretion by the liver can be evaluated; 4. Provide a pathway for cholangiography. However, placing external biliary drainage may also pose certain risks, including increasing surgical procedures, stent detachment causing biliary fistula, and increasing the risk of infection.

This study aims to observe the effect of placing external biliary drainage stents on biliary stricture after liver transplantation in children. The aim is to evaluate the preventive effect of external biliary drainage stents on biliary intestinal anastomotic stenosis after liver transplantation in children, and to provide evidence-based evidence for reducing biliary complications in children.

ELIGIBILITY:
Inclusion Criteria:

1. The patient underwent liver transplantation surgery at the First Affiliated Hospital of Zhejiang University School of Medicine;
2. Age ≤ 6 years old;
3. First liver transplantation;
4. Willing to sign an informed consent form.

Exclusion Criteria:

- Existence of mental illnesses that can affect cognition and coordination.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients need liver transplantation
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
duct-jejunum anastomotic stoma stricture | one year
  number of participants with duct-jejunum anastomotic stoma stricture after liver transplantation

SECONDARY OUTCOMES:
biliary tract infection | one year
  number of participants with biliary tract infection after liver transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China